CLINICAL TRIAL: NCT03063060
Title: The Impact of Vitamin D Deficiency on Hypocalcaemia Following Total Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Ahud Sternberg, Chairman of ethics board, Hillel Yaffe Medical Center
Other Study IDs: 0014-17
Record Dates: First submitted 2017-01-25; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Hypocalcemia; Vitamin D Deficiency
MeSH Terms: conditions — Hypocalcemia; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- total thyroidectomy: patients who underwent total thyroidectomy with available vitamin D levels before surgery, as well as pre and post-operative PTH and calcium levels.
  Interventions: Other: vitamin D levels and Calcium levels examination

INTERVENTIONS:
Other: vitamin D levels and Calcium levels examination — observational

SUMMARY:
Post-operative hypocalcaemia following total thyroidectomy is a well-known complication and becoming a major area of research.

Many factors are assumed to increase the incidence of post-thyroidectomy hypocalcaemia, but the impact of vitamin D deficiency remains uncertain.

Since results so far were inconclusive, the goal in this study is to significantly determine the relation between those two factors.

This study is the first to deal with this issue through patients who underwent total thyroidectomy that was performed by the same surgeon and the same surgical technique.

A retrospective evaluation study of patients who underwent total thyroidectomy at the head and neck unit of the Otorhinolaryngology department at our institution between January 2013 and October 2016.

A total number of 60 patients underwent total thyroidectomy with available vitamin D levels before surgery, as well as pre and post-operative PTH and calcium levels.

Pre-operative vitamin D and PTH levels were checked within a maximum of one month duration before surgery.

All patients were operated by the same surgeon -Dr. Galit Avior-, with the same surgical technique.

The study involves access to the patients files and admission reports. In addition the investigators would like to be able to call the patients in order to ask them whether Vitamin D deficiency was corrected or not before their surgery, and If it was corrected then when exactly.

DETAILED DESCRIPTION:
Background Post-operative hypocalcaemia following total thyroidectomy is a well-known complication and becoming a major area of research.

Many factors are assumed to increase the incidence of post-thyroidectomy hypocalcaemia, but the impact of vitamin D deficiency remains uncertain.

Vitamin D deficiency is known to be one of the most common medical conditions in the world.. Serum calcium is mainly regulated by parathyroid hormone (PTH) and vitamin D, therefore demonstration of a correlation between preoperative vitamin D levels and the occurrence of post thyroidectomy hypocalcaemia may reveal an easily correctable factor.

Recently, few studies have investigated whether preoperative vitamin D levels have any effect on post thyroidectomy hypocalcaemia. Some of them showed that patients with vitamin D deficiency were more likely to develop postoperative hypocalcaemia. In addition a significant decrease in postoperative hypocalcemia was shown in patients who received supplementation of vitamin D regardless of their vitamin D status, while others found no relationship between preoperative vitamin D concentrations and postoperative hypocalcaemia .

Since results so far were inconclusive, the goal in this study is to significantly determine the relation between those two factors.

This study is the first to deal with this issue through patients who underwent total thyroidectomy that was performed by the same surgeon and the same surgical technique.

Study objective

1. To identify a correlation between pre-operative vitamin D deficiency and the occurrence of hypocalcaemia following total thyroidectomy.
2. To determine wether the correction of vitamin D levels prior to the surgery was able to prevent post surgery hypocalcaemia.

Study design A retrospective evaluation study of patients who underwent total thyroidectomy at the head and neck unit of the Otorhinolaryngology department at our institution between January 2013 and October 2016.

A total number of 60 patients underwent total thyroidectomy with available vitamin D levels before surgery, as well as pre and post-operative PTH and calcium levels.

Pre-operative vitamin D and PTH levels were checked within a maximum of one month duration before surgery.

All patients were operated by the same surgeon -Dr. Galit Avior-, with the same surgical technique.

Methods:

The study involves access to the patients files and admission reports. In addition the investigators would like to be able to call the patients in order to ask them whether Vitamin D deficiency was corrected or not before their surgery, and If it was corrected then when exactly.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years.
* Both males and females.
* Patients who underwent total thyroidectomy.
* Documented 25-hydroxyvitamin D level preoperatively.
* Documented calcium levels pre and postoperatively.
* Documented PTH levels pre and postoperatively.

Exclusion Criteria:

* Patients with either hypocalcaemia or hypercalcemia before surgery.
* Patients with Grave's disease.
* Patients with renal, lung or bone cancer.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total number of 60 patients underwent total thyroidectomy with available vitamin D levels before surgery, as well as pre and post-operative PTH and calcium levels.
  Pre-operative vitamin D and PTH levels were checked within a maximum of one month duration before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin D levels | pre- operative vitamin D levels 1 month prior to surgery
  ng/ml
Calcium levels | post operative Ca levels at the day of the surgery
  mg/dl
Calcium levels | post operative Ca levels 1 day after the surgery
  mg/dl

IPD SHARING:
Plan to Share IPD: Undecided